CLINICAL TRIAL: NCT03639142
Title: Dried Plums (Prunes) vs. Polyethylene Glycol 4000 for Treatment of Functional Constipation in Children - Randomised Controlled Trial
Brief Title: Dried Plums (Prunes) vs. Polyethylene Glycol 4000 for Treatment of Functional Constipation in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Piotr Dziechciarz, MD, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1/2018
Record Dates: First submitted 2018-08-14; First posted 2018-08-20 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Functional Constipation
Keywords: constipation, prunes, children
MeSH Terms: conditions — Constipation | interventions — polyethylene glycol 4000

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plum group (Experimental): Children will receive plums at dose 3,5g/kg/d as an oral treatment for constipation.
  Interventions: Other: Prunus domestica
- Polyethylene glycol group (Active Comparator): Children will receive PEG at dose 0,5g/kg/d as an oral treatment for constipation.
  Interventions: Drug: Polyethylene Glycol 4000

INTERVENTIONS:
Other: Prunus domestica — Patients will receive prunes at dose 3,5 g/kg/d (max.100mg/day) in three portions a day, for 4 weeks (amount of prescribed prunes will be calibrated with the weight that child ought to have on WHO growth charts at 50th percentile). Prunes should be introduced every day in three meals. Prunes can be chopped or grinded before eating them. They can be eaten alone or child may eat them as a part of bigger meal (which is preferred version). Prunes can be introduced with yogurt, cereals, nuts and seeds as a morning meal.
  Arms: Plum group
Drug: Polyethylene Glycol 4000 — Patients will receive PEG at dose 0,5 g/kg/d once daily orally, for 4 weeks.
  Arms: Polyethylene glycol group

SUMMARY:
Children with functional constipation according to the Rome IV criteria will be randomly assigned to receive prunes at dose 3.5 g/kg/d (prune group) or Polyethylene Glycol 4000 (PEG group) at dose 0.5 g/kg/d for 4 weeks. Before treatment children with impaction will receive PEG 4000 at the dose 1.5 g/kg for 3-5 consecutive days. The primary outcome measure will be treatment success, defined as ≥3 BM per week with no fecal soiling during last week of the intervention.

DETAILED DESCRIPTION:
We will conduct a randomized open-label trial at the Department of Paediatrics of the Medical University of Warsaw. The trial will be initiated by the investigators and conducted independently of any commercial entities. The aim will be to assess the effectiveness of dried prunes in the management of functional constipation in children in comparison to PEG 4000. Patients will be included into our study when functional constipation will be diagnosed according to ROME IV criteria. Those patients which will meet inclusion criteria will be assigned randomly to receive prunes at dose 3,5 g/kg/d in three portions a day, for 4 weeks (amount of prescribed prunes will be calibrated with the weight that child ought to have on WHO growth charts at 50th percentile) or PEG 4000 at dose 0,5 g/kg/d once daily orally, for 4 weeks. Parents of the children allocated to the prunes group will receive written information from dietician how to introduce prunes into child's diet (i.e. prunes should be introduced every day in three meals; prunes can be chopped or grinded before eating them; prunes can be eaten alone or child may eat them as a part of bigger meal (which is prefered version); prunes can be introduced with yoghurt, cereals, nuts and seeds as a morning meal). All patients will be asked to discontinue any laxatives if they used them previously. In case of rectal impaction noted on physical examination, PEG 4000 at dose of 1.5 g/kg for 3-5 consecutive days will be recommended. All subjects parents will receive a stool diary to record the frequency of bowel movements; stool consistency according to Bristol Stool Form Scale (which refers to 7 pictures of different forms of stool; 1 for hard lumps to 7 for watery stools); frequency of episodes of fecal soiling, pain during defecation, or abdominal pain or flatulence; use of additional laxative treatment; and adverse effects during the 4 weeks of the intervention. All patients or their parents (if child is too young) will be asked to write down selfreported 3 day food diaries on non-consecutive days, 2 d during the week and 1 d during the weekend to assess fiber intake during the study period .. All patients will be informed of rescue therapy -when there will be no defecation for 3 consecutive days during ongoing trail, PEG 4000 will be allowed at the dose of 1.5 g/kg/d until the child will pass a stool.

During the study period, every week investigator will call the patients parents to assess compliance with the study protocol.

Second visit will take place at the end of the trial (4th week). During this visit, investigators will collect stool diaries. Prunes used in the study will be purchased by parents of the children. It will be advised for parents to buy prunes under the trade mark of "Makar" in order to avoid product composition variability bias. Choice of the trade mark was taken considering the price of a product.

This study is designed as a randomized, open label controlled trial with 1:1 allocation. In order to obtain comparable groups, block randomisation will be performed (each block will contain four patients: two in the intervention group and two in the control group). The randomisation list will be generated using the statistical program StatsDirect by an independent person and will be kept by a staff member not involved in the trial.

Based on available data in the literature, we assume that a clinically significant difference in the effectiveness is 15%. To detect such a difference between the study groups with a power of 80% and alpha of 5%, a sample of 100 children is needed. Assuming approximately 10% loss to follow-up, we aim to recruit a total of 110 children for this study.

The Ethical Committee of the Medical University of Warsaw will be asked for approval for the study before recruitment commenced. Any modifications to the protocol that may affect the conduct of the study will be presented to the Ethical Committee. Verbal and written information regarding informed consent will be presented to the caregivers.

All analysis will be conducted on an intention-to-treat basis, including all patients in the groups to which they are randomized for whom outcomes are available (including drop-outs and withdrawals). Descriptive statistics will be used to summarize baseline characteristics. The Student t test will be used to compare mean values of continuous variables for approximating a normal distribution. For non normally distributed variables, the Mann-Whitney U test will be used. The chi-square or Fisher exact test will be used, when appropriate, to compare percentages. For continuous outcomes, differences in means or differences in medians (depending on the distribution of the data), and for dichotomous outcomes, the RR and number needed to treat, all with a 95% CI, will be calculated. The difference between study groups will be considered significant when the 95% CI for RR does not include 1.0, or when the 95% CI for MD does not include 0. All statistical tests will be 2-tailed and performed at the 5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

* children with constipation diagnosed with ROME IV criteria

Exclusion Criteria:

* diagnosis of irritable bowel syndrome, mental retardation, endocrine disease (eg, Hyperthyroidism), an organic cause of defecation disorders (eg, Hirshsprung disease, spinal anomalies, anorectal pathology, a history of gastrointestinal surgery), functional nonretentive fecal incontinence, or intake of medications influencing gastrointestinal motility

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be treatment success | up to 4 weeks
  ≥3 spontaneous stools per week, without episodes of fecal soiling (in toilet-trained children), in the last week of the intervention (week 4).

SECONDARY OUTCOMES:
stool consistency (according to the Bristol Stool Form Scale) during whole study period | up to 4 weeks
  Scale ranges from 1 to 7 where types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid, 5 tending towards diarrhoea, and 6 and 7 indicate diarrhoea.
frequency of defecation per week | up to 4 weeks
frequency of fecal soiling per week | up to 4 weeks
frequency of pain during defecation per week | up to 4 weeks
frequency of abdominal pain or flatulence per week | up to 4 weeks
need for intake of additional laxative treatment during whole study period | up to 4 weeks
adverse events | up to 4 weeks

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Attaluri A, Donahoe R, Valestin J, Brown K, Rao SS. Randomised clinical trial: dried plums (prunes) vs. psyllium for constipation. Aliment Pharmacol Ther. 2011 Apr;33(7):822-8. doi: 10.1111/j.1365-2036.2011.04594.x. Epub 2011 Feb 15. PMID 21323688
- [Background] Benninga MA, Faure C, Hyman PE, St James Roberts I, Schechter NL, Nurko S. Childhood Functional Gastrointestinal Disorders: Neonate/Toddler. Gastroenterology. 2016 Feb 15:S0016-5085(16)00182-7. doi: 10.1053/j.gastro.2016.02.016. Online ahead of print. PMID 27144631
- [Background] Chmielewska A, Horvath A, Dziechciarz P, Szajewska H. Glucomannan is not effective for the treatment of functional constipation in children: a double-blind, placebo-controlled, randomized trial. Clin Nutr. 2011 Aug;30(4):462-8. doi: 10.1016/j.clnu.2011.01.012. Epub 2011 Feb 12. PMID 21320737
- [Background] Dehghani SM, Kulouee N, Honar N, Imanieh MH, Haghighat M, Javaherizadeh H. Clinical Manifestations among Children with Chronic Functional Constipation. Middle East J Dig Dis. 2015 Jan;7(1):31-5. PMID 25628851
- [Background] Dziechciarz P, Horvath A, Szajewska H. Polyethylene glycol 4000 for treatment of functional constipation in children. J Pediatr Gastroenterol Nutr. 2015 Jan;60(1):65-8. doi: 10.1097/MPG.0000000000000543. PMID 25162362
- [Background] Horvath A, Dziechciarz P, Szajewska H. Glucomannan for abdominal pain-related functional gastrointestinal disorders in children: a randomized trial. World J Gastroenterol. 2013 May 28;19(20):3062-8. doi: 10.3748/wjg.v19.i20.3062. PMID 23716985
- [Background] Koppen IJ, Nurko S, Saps M, Di Lorenzo C, Benninga MA. The pediatric Rome IV criteria: what's new? Expert Rev Gastroenterol Hepatol. 2017 Mar;11(3):193-201. doi: 10.1080/17474124.2017.1282820. Epub 2017 Jan 24. PMID 28092724
- [Background] Lever E, Cole J, Scott SM, Emery PW, Whelan K. Systematic review: the effect of prunes on gastrointestinal function. Aliment Pharmacol Ther. 2014 Oct;40(7):750-8. doi: 10.1111/apt.12913. Epub 2014 Aug 11. PMID 25109788
- [Background] Mugie SM, Benninga MA, Di Lorenzo C. Epidemiology of constipation in children and adults: a systematic review. Best Pract Res Clin Gastroenterol. 2011 Feb;25(1):3-18. doi: 10.1016/j.bpg.2010.12.010. PMID 21382575
- [Background] Tabbers MM, DiLorenzo C, Berger MY, Faure C, Langendam MW, Nurko S, Staiano A, Vandenplas Y, Benninga MA; European Society for Pediatric Gastroenterology, Hepatology, and Nutrition; North American Society for Pediatric Gastroenterology. Evaluation and treatment of functional constipation in infants and children: evidence-based recommendations from ESPGHAN and NASPGHAN. J Pediatr Gastroenterol Nutr. 2014 Feb;58(2):258-74. doi: 10.1097/MPG.0000000000000266. PMID 24345831
- [Background] Zeevenhooven J, Koppen IJ, Benninga MA. The New Rome IV Criteria for Functional Gastrointestinal Disorders in Infants and Toddlers. Pediatr Gastroenterol Hepatol Nutr. 2017 Mar;20(1):1-13. doi: 10.5223/pghn.2017.20.1.1. Epub 2017 Mar 27. PMID 28401050